CLINICAL TRIAL: NCT01262859
Title: Pilot Study of Induction Docetaxel, Cisplatin, Cetuximab and Bevacizumab (TPE-A) Followed by Concurrent Radiation, Cisplatin, Cetuximab and Bevacizumab (XPE-A) in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Pilot Study for Locally Advanced Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI relocated to another institution. No subjects went on treatment.
Sponsor: University of Pittsburgh (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Athanassios Argiris, MD, UPCI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-039; UPCI 09-039 (Other: University of Pittsburgh Cancer Institute identifier)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Intervention (Experimental): Induction therapy consists of 3 cycles of bevacizumab 15mg/kg on day 1, cetuximab weekly days 1,8,15 (loading dose of cetuximab 400mg/m2 on cycle 1, day 1, then 250 mg/m2 on all subsequent administrations), cisplatin 75mg/m2 on day 1, docetaxel 75mg/m2 on day 1, repeated every 21 days. After 3 cycles of induction therapy, patients will receive standard radiation 70-74 Gy/ 200 cGy/ daily, 5 days/ week with concurrent weekly cisplatin 30mg/m2, cetuximab 250mg/m2 and bevacizumab 15mg/kg every 3 weeks x 3. There is optional surgery for non-responders in the primary (stable disease) after TPE-A.
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — Bevacizumab, 15 mg/kg IV over 30 minutes (if this infusion rate was well tolerated), every 3 weeks until completion of radiation The initial dose will be delivered over 90+/-15 minutes. If the first infusion is tolerated without infusion associated adverse events (fever and/or chills), the second infusion may be delivered over 60+/-10 minutes. If the 60 minute infusion is well tolerated, all subsequent infusions may be delivered over 30+/-10 minutes.
  Other Names: Avastin

SUMMARY:
Induction chemotherapy is gaining momentum in the management of locally advanced squamous cell carcinoma of the head and neck (SCCHN). The combination of docetaxel, cisplatin, and 5-FU (TPF) was superior compared with PF in a Phase III clinical trials73,74. We have completed a Phase II clinical trial that showed that docetaxel, cisplatin, and cetuximab (TPE) is highly active and well tolerated as induction chemotherapy in SCCHN (Argiris et al. ASCO 2008; A6002). Preliminary survival results are very encouraging. 39 patients were enrolled and with median follow up 26 months the 2-year PFS was 70% and the 2-year OS 84%.The combination of chemotherapy plus cetuximab is already a standard treatment in recurrent or metastatic SCCHN47. Therefore, TPE can be used as the platform for the addition of novel agents.

EGFR and VEGF are among the most important and validated molecular targets in cancer therapy. The incorporation of novel targeted therapies to chemotherapy and radiotherapy is of particular interest in head and neck cancer, and may improve efficacy without significantly increasing toxicity. A Phase III trial of carboplatin/paclitaxel/bevacizumab with or without cetuximab in advanced NSCLC has been proposed by SWOG. Bevacizumab is currently being investigated in SCCHN with promising results. A Phase II study investigating the combination of pemetrexed and bevacizumab (UPCI 05-002) as well as a Phase II trial of cetuximab and bevacizumab (UPCI 05-087) in recurrent or metastatic SCCHN are ongoing at the University of Pittsburgh with encouraging results (ASCO 2008 and ASCO 2009). In this study, 32 have been already enrolled. There was only 1 patient with grade 3 hemorrhage. The objective response rate is 20%, the median PFS 2.8 months and the median OS 8.1 months.

In order to further improve the efficacy of TPE and the rate of complete responses we propose to add bevacizumab to the TPE followed by XPE regimen we developed at the University of Pittsburgh. Due to non-overlapping toxicities and based on our prior experience we anticipate that the regimen will be well tolerated. Moreover, we plan to obtain tumor biopsies and blood samples in the first cycle and evaluate the modulation of biomarkers post combination therapy. Data from induction with TPE (presented at ASCO 2009) indicate the potential significance of cytokine levels in patient outcome. Also, we will evaluate the feasibility of subsequent concurrent radiation, cisplatin, cetuximab and bevacizumab. Patients with stable disease in the primary could be considered candidates to surgical resection at the discretion of their physician, if the tumor is resectable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AJCC 6th edition stage III-IVB head and neck cancer, all sites, including unknown primary tumors.
* Prior to entry in the study the resectability and alternative treatment options for each patient will be determined by a team composed of an Ear, Nose, and Throat Surgeon, a Radiation Oncologist and a Medical Oncologist. Stage determination, optimal local treatment, and its timing according to this protocol will be determined at this evaluation. The unequivocal demonstration of distant metastasis (M1) confers ineligibility.
* Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas, or WHO types I-III of the nasopharynx.
* Unidimensionally measurable disease is required (RECIST 1.1).
* No prior chemotherapy, biologic/molecular targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer.
* Prior surgical therapy will consist only of incisional or excisional biopsy, and organ sparing procedures such as debulking of airway compromising tumors or neck dissection in a patient with an existing primary tumor. Any non-biopsy procedure must have taken place > 4 weeks but < 3 months of initiating protocol treatment.
* ECOG performance status 0-1.
* Age of at least 18 years.
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* All patients should have their tumor tissue tested for HPV and will consent to have available archival tumor samples, unstained slides or blocks from previous diagnostic or therapeutic procedures submitted for correlative studies, including assessment of target molecules EGFR, VEGF and related biomarkers. Also, patients must agree to submit blood samples for correlative studies at least at baseline.
* Absolute neutrophil count equal to or greater than 1500/µl, Platelet count equal to or greater than 100,000/µl
* Creatinine clearance 60 ml/min or higher calculated using the Cockcroft-Gault formula:

Calculated Creatinine Clearance = (140-age) X actual body wt.(kg) 72 X serum creatinine Multiply this number by 0.85 if the patient is female

* Total bilirubin within normal limits and AST/ALT less than 3 times the upper limit of normal.
* Urine to protein to creatinine (UPC) ratio should be <1.0 at screening

NOTE: UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1gm. UPC ratio is calculated using one of the following formula:

* [urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/DI
* [(urine protein) × 0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

  * Patients with a prior history of squamous cell or basal carcinoma of the skin or in situ cervical cancer must have been curatively treated. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post diagnosis.
  * Patients may not be receiving any other investigational agents.

Exclusion Criteria:

* History of severe allergic reactions attributed to docetaxel or compounds of similar chemical or biologic composition to docetaxel, or other drugs formulated with polysorbate 80.
* Prior severe infusion reaction to a monoclonal antibody or known hypersensitivity to any component of bevacizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study
* No patients with significant baseline sensory or motor neurologic deficits (> grade I neuropathy) will be treated on this study.
* Because patients with immune deficiency are at increased risk of lethal Infections when treated with marrow-suppressive therapy, HIV-positive patients are excluded from the study. Appropriate studies will be undertaken in patients with HIV and those receiving combination anti- retroviral therapies when indicated.
* Patients with HPV positive tumors
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix F)
* History of myocardial infarction or unstable angina within 12 months prior to Day 1
* No history of stroke or transient ischemic attack within 6 months prior to Day 1
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (equal to or greater than 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Patients should not be on therapeutic anticoagulation therapy (prophylactic use of warfarin 1mg per day is allowed) and INR should be <1.5 at registration
* The use of anti-platelet agents (e.g. dipyridamole (Persatine), ticlopidine (Ticlid), clopidogrel (Plavix)) is allowed only if patient is not receiving aspirin or NSAID's known to inhibit platelet function.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Pregnant or breast-feeding women will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Response rate | 10 years
  To evaluate the rate of complete responses with induction with cisplatin, docetaxel, cetuximab and bevacizumab (TPE-A) in patients with locally advanced head and neck cancer.

SECONDARY OUTCOMES:
Serum Correlatives | 10 years
  To evaluate serum cytokines and to correlate with complete response rate post induction therapy.
Biomarkers | 10 years
  To collect tumor tissue from pretreatment and post-treament (optional) biopsies for biomarker studies on tumor tissue. We plan to investigate a panel of EGFR and angiogenesis biomarkers on Tissue Microarrays (TMAs).
Toxicity | 10 years
  To evaluate the toxicities associated with induction TPE-A and subsequent concurrent radiation, cispaltin, cetuximab and bevacizumab (XPE-A).
Response rate and progression-free survival | 10 years
  To evaluate the objective response rate post XPE-A, and the progression- free survival and overall survival and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States